CLINICAL TRIAL: NCT04341545
Title: Randomized Controlled Trial on Use of Letrozole in the Medical Management of Tubal Ectopic Pregnancies
Brief Title: Letrozole in Tubal Ectopic Pregnancy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Pamela Youde Nethersole Eastern Hospital, Hong Kong (Unknown); Queen Elizabeth Hospital, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Evelyn Wong, Associate consultant, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 20-005
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Tubal Pregnancy
Keywords: Tubal ectopic pregnancy; Methotrexate; Letrozole
MeSH Terms: conditions — Pregnancy, Tubal | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either receive letrozole or placebo capsules.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The identical looking placebo will be given. A computer generated sequence will be created. The sequence will be sealed in consecutively concealed opaque envelopes. Both the participant/ care provider/ investigator and outcomes assessor will blinded to the group assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): Participants will be given letrozole 10mg daily for one week after standard medical management for tubal ectopic pregnancy by methotrexate injection. Subsequently they will receive the standard management for medical management of tubal ectopic prengnacies.
  Interventions: Drug: Letrozole tablets
- Placebo (Placebo Comparator): Participants will be given identical looking placebo for one week and receive the same standard management for medical management of tubal ectopic pregnancies.
  Interventions: Other: Placebos

INTERVENTIONS:
Other: Placebos — Placebo 4 tablets a day for one week.
  Arms: Placebo
Drug: Letrozole tablets — Letrozole 10mg daily for one week.
  Other Names: Letrozole
  Arms: Letrozole

SUMMARY:
This is a multi-centred randomized controlled trial on the addition of letrozole in the medical management of tubal ectopic pregnancies.

Tubal ectopic pregnancies are abnormal pregnancies in the Fallopian tube, rather than in the womb. They occurred in around 1-2% of all pregnancies. Methotrexate (MTX) given by the intramuscular route i.e. systemic, a commonly used drug for cancer , was a widely used alternative for management for unruptured tubal ectopic pregnancies and was recommended as first line treatment for selected women.

Letrozole, aromatase inhibitor, can suppose oestradiol level. Combination of letrozole with misprostol has shown to improve the complete abortion rate in miscarriage. As a result, addition of letrozole may cause a higher success rate in the medical treatment of ectopic pregnancy.

As the evidence of combination of MTX and letrozole in tubal ectopic pregnancies is not available, the objective of the present study is to evaluate the efficacy of combination of MTX and letrozole compared to MTX alone in women with tubal ectopic pregnancies.

DETAILED DESCRIPTION:
Tubal ectopic pregnancies occur in around 1-2% of all pregnancies. Traditionally, surgery with salpingectomy was the mainstay of treatment; however, it comes with anaesthetic and operatives risks in addition to an increased cost for operative procedures. In recent years, systemic methotrexate (MTX), a dihydrofolate reductase inhibitor, has been a widely used alternative for management for unruptured tubal ectopic pregnancies. The success rate of systemic MTX at a doses of 50mg/m2 body surface area is around 70% which ranges from 65 to 95%, depending greatly on the level of human chorionic gonadotrophin (hCG), the size of adnexal mass and presence of fetal heart pulsation.

Use of systemic MTX as the first-line management has been proposed for women with unruptured ectopic pregnancy where the adnexal mass is smaller than 35mm, serum hCG level is less than 5000 IU/l and fetal heartbeat is absent.

Letrozole is a third generation non-steroidal reversible aromatase inhibitor. It can suppress oestradiol level up to 95% to 99% after administration according to pharmacodynamics and pharmacokinetics studies. Oestrogen is important in the support of early pregnancy, other than progesterone with well-known pivotal effect on the maintenance of early pregnancy.

Animal studies showed the combination of mifepristone and letrozole worked synergistically and induced almost 100% termination of pregnancies in rats. Letrozole induced 50% miscarriage rate in pregnant baboons. Letrozole combined with vaginal misoprostol regimen was associated with a higher complete abortion rate than misoprostol alone in pregnancies up to 63 days.

The use of letrozole in ectopic pregnancy has never been explored. It is hypothesized that letrozole can suppress serum oestradiol level, which in turn, may cause failure of pregnancy in ectopic pregnancy. The aim of this study is to investigate the clinical effectiveness of letrozole in addition to MTX in the medical treatment of ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of heterogenous adnexal mass on USG suggestive of tubal ectopic pregnancy with hCG level >=1500 IU/L and <= 5000 IU/L
* Absence of fetal heart pulsation
* Mean diameter of adnexal mass <= 3.5cm
* Haemodynamically stable
* No significant abdominal pain

Exclusion Criteria:

* Presence of significant amount of free fluid in pelvis
* Allergic to MTX
* Deranged liver function test (AST/ ALT or GGT >= 2 upper limit of normal)
* Deranged renal function test (eGFR <= 45ml/min)
* Heterotopic pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ectopic pregnancies studied
Enrollment: 214 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 2 months
  Proportion of women with treatment success defined as normalization of serum hCG level <10IU/L without additional medical or surgical intervention

SECONDARY OUTCOMES:
hCG normalization duration | 2 months
  Duration of time until hCG normalization measured in days
Number of participants experienced side effects | 2 months
  Side effects after letrozole
Duration of hospitalization | 2 months
  Duration of hospitalization
Participant satisfaction: proportion of women who would recommend this treatment to a friend | 2 months
  Treatment satisfaction measured as proportion of women who would recommend this treatment to a friend

CONTACTS AND LOCATIONS:
Overall Officials: Ernest H.Y. Ng, MD, Study Director — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Other researchers may contact the chief investigator for the request of individual participant data.

REFERENCES:
- [Background] Panelli DM, Phillips CH, Brady PC. Incidence, diagnosis and management of tubal and nontubal ectopic pregnancies: a review. Fertil Res Pract. 2015 Oct 15;1:15. doi: 10.1186/s40738-015-0008-z. eCollection 2015. PMID 28620520
- [Background] Diagnosis and Management of Ectopic Pregnancy: Green-top Guideline No. 21. BJOG. 2016 Dec;123(13):e15-e55. doi: 10.1111/1471-0528.14189. Epub 2016 Nov 3. No abstract available. PMID 27813249
- [Background] Odejinmi F, Huff KO, Oliver R. Individualisation of intervention for tubal ectopic pregnancy: historical perspectives and the modern evidence based management of ectopic pregnancy. Eur J Obstet Gynecol Reprod Biol. 2017 Mar;210:69-75. doi: 10.1016/j.ejogrb.2016.10.037. Epub 2016 Oct 29. PMID 27940397
- [Background] National Collaborating Centre for Ws, Children's H. National Institute for Health and Clinical Excellence: Guidance. Ectopic Pregnancy and Miscarriage: Diagnosis and Initial Management in Early Pregnancy of Ectopic Pregnancy and Miscarriage. London: Rcog National Collaborating Centre for Women's and Children's Health.; 2012.
- [Background] Shi L, Shi SQ, Given RL, von Hertzen H, Garfield RE. Synergistic effects of antiprogestins and iNOS or aromatase inhibitors on establishment and maintenance of pregnancy. Steroids. 2003 Nov;68(10-13):1077-84. doi: 10.1016/j.steroids.2003.09.002. PMID 14668001
- [Background] Albrecht ED, Aberdeen GW, Pepe GJ. The role of estrogen in the maintenance of primate pregnancy. Am J Obstet Gynecol. 2000 Feb;182(2):432-8. doi: 10.1016/s0002-9378(00)70235-3. PMID 10694348
- [Background] Lee VCY, Ng EHY, Yeung WSB, Ho PC. Misoprostol with or without letrozole pretreatment for termination of pregnancy: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):317-323. doi: 10.1097/AOG.0b013e3182073fbf. PMID 21252745
- [Background] Lee VC, Tang OS, Ng EH, Yeung WS, Ho PC. A pilot study on the use of letrozole with either misoprostol or mifepristone for termination of pregnancy up to 63 days. Contraception. 2011 Jan;83(1):62-7. doi: 10.1016/j.contraception.2010.05.014. Epub 2010 Jun 23. PMID 21134505